CLINICAL TRIAL: NCT03026582
Title: Intestinal Ultrasound Role in the Management of Pediatric Inflammatory Bowel Disease: A Prospective Longitudinal Cohort Study
Brief Title: Intestinal Ultrasound in Pediatric Inflammatory Bowel Disease
Acronym: SPIBDUS
Status: Completed | Type: Observational
Sponsor: Schneider Children's Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Amit Assa, Head of IBD program, Schneider Children's Medical Center, Israel
Other Study IDs: SchneiderCMCIsrael
Record Dates: First submitted 2017-01-16; First posted 2017-01-20 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Intestinal ultra-sound monitoring — Children diagnosed with either CD or UC will be enrolled at diagnosis or at any time point during follow-up. Patients' characteristics will be retrieved from their medical files including demographic details, disease phenotype, endoscopic and radiologic variables, anthropometric measures, laboratory evaluation, complication and therapeutic regimens. At enrollment and every 3 months for a total period of 2 years all patients will perform intestinal US during regular clinic visits. All other measures including laboratory exams, anthropometric measurements and disease activity indices (either PCDAI for CD or PUCAI for UC) will be performed as part of standard of care.

SUMMARY:
Objectives: To assess the predictive value of IUS in children with IBD.

Design: A prospective longitudinal cohort study.

Setting: Institute of Gastroenterology, Nutrition and Liver Diseases, Schneider Children's Hospital.

Participants: Children 2 years to 17 years (up to 200 patients) who have been diagnosed with either CD or UC.

Main outcome measures: The changes in bowel wall thickness, assessed by IUS, during 2-year follow-up according to therapeutic regimen.

Secondary outcome measures: Correlation of sonographic measures to clinical disease indices, serum inflammatory and other laboratory markers, fecal calprotectin, endoscopic and other radiologic measures performed as part of routine care.

DETAILED DESCRIPTION:
Hypothesis:

The investigators hypothesize that bowel wall thickness as measured routinely by IUS has a role in predicting short- and long-term disease outcomes such as flares, hospitalizations, treatment escalation and surgery.

Objectives:

Primary Objectives:

To assess the changes in bowel wall thickness, assessed by IUS, during 2-year follow-up, according to therapeutic regimen and to evaluate its predictive significance on disease outcomes (flares, hospitalizations, treatment escalation and surgery).

Secondary Objective: To evaluate the correlation of sonographic measures to clinical disease indices, serum inflammatory and other laboratory markers, fecal calprotectin, endoscopic and other radiologic measures performed as part of routine care.

Methods:

* Design: A prospective longitudinal cohort study.
* Patients: Children at age 2 year to 17 years diagnosed with IBD.

Intervention:

Children diagnosed with either CD or UC under follow-up at the Institute of Gastroenterology, Nutrition and Liver Diseases, Schneider Children's Hospital, will be enrolled. Patients can be enrolled at diagnosis or at any time point during follow-up. Patients' characteristics will be retrieved from their medical files including demographic details, disease phenotype, endoscopic and radiologic variables, anthropometric measures, laboratory evaluation, complication and therapeutic regimens. At enrollment and every 3 months for a total period of 2 years all patients will perform IUS during regular clinic visits. All other measures including laboratory exams, anthropometric measurements and disease activity indices (either wPCDAI for CD or PUCAI for UC) will be performed as part of standard of care and not for the purpose of the study. If endoscopic evaluation or an MRE are necessary according to the treating physician discretion for assessment of disease activity, these will not be performed as part of the study but the results will be recorded and included in the data analysis.

Data analysis:

Data will be analyzed using SPSS (version 23.0, SPSS, Inc., Armonk, NY, USA) and r-project version 3.1.1. Continues variables will be presented as either mean±SD or median with interquartile range (IQR) depending on the data approximation to normal distribution. Agreement between IUS and MRE (when available) will be assessed using Bland-Altman plot and Concurrent Validity quantified by correlation coefficient and concordance correlation coefficient. Associations of therapeutic intervention and other variables with outcome measures will be examined using repeated measures ANOVA. p-values <0.05 is considered significant.

Sample size:

All pediatric IBD patients at Schneider Children's Hospital, fulfilling the inclusion criteria are eligible for the study. For assessment of therapeutic interventions of IUS the investigators will use mixed model ANOVA. Sample size was calculated for repeated measures ANOVA with in-between interactions. Assuming effect size F 0.25 (or partial η2=0.06), an alpha of 5% and statistical power of 80% and a correlation of 0.5, the investigators will need at least 34 CD patients and 34 UC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of IBD
2. Age: 2- 17 years (inclusive)
3. Informed consent

Exclusion Criteria:

1. Pregnancy
2. Morbid obesity

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 2 years to 17 years who have been diagnosed at the Schneider Children's Hospital with either Crohn's disease or ulcerative colitis.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change in bowel wall thickness according to therapeutic regimen | Two years

SECONDARY OUTCOMES:
Change in bowel wall thickness in comparison to inflammatory markers | Two years
Change in bowel wall thickness in comparison to fecal calprotectin | Two years
Change in bowel wall thickness in comparison to pediatric Crohn's disease severity index in Crohn's disease | Two years
Change in bowel wall thickness in comparison to pediatric ulcerative colitis activity index in ulcerative colitis | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Amit Assa, Principal Investigator — Schneider Children's Medical Center, Israel
Locations (1):
- Schenider Children's Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No